CLINICAL TRIAL: NCT04789473
Title: Gestational Diabetes Genetic and Socioeconomic Risk Study OneinSeven Gestational Diabetes Genetic and Socioeconomic Risk Study
Brief Title: OneinSeven Gestational Diabetes Genetic and Socioeconomic Risk Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prenome (Industry)
Responsible Party: Sponsor
Other Study IDs: PRE001
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Gestational Diabetes; Pregnancy Complications; Pregnancy Related; Genetic Predisposition; Risk Reduction
Keywords: Gestational Diabetes; Polygenic Risk Score; Genomics
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy Complications; Genetic Predisposition to Disease; Risk Reduction Behavior; Genetic Risk Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva specimens used for DNA collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Normal Glycemic Pregnancy: Cohort of control adults who are currently pregnant or have been pregnant within the last year, but were not diagnosed with gestational diabetes.
  Interventions: Genetic: Polygenic Risk Score Generation
- Gestational Diabetic Cohort: Cohort of adults who are currently pregnant or have been pregnant within the last year, but were diagnosed with gestational diabetes.
  Interventions: Genetic: Polygenic Risk Score Generation

INTERVENTIONS:
Genetic: Polygenic Risk Score Generation — PRS will be calculated for gestational diabetes risk using both cohorts, participants wont have results returned to them during the study.

SUMMARY:
The objective of the Gestational Diabetes Genetic Socioeconomic Risk Study is to generate genome wide association study data (GWAS) to calculate polygenic risk scores (PRS) for the development of gestational diabetes in pregnant women. Oshun Medical's GWAS study will be conducted by collecting DNA samples alongside medical and socioeconomic data and applying data science methodology to generate a polygenic risk score algorithm for gestational diabetes. Our hypothesis is that key genetic variants linked to gestational diabetes will be identified, and sociodemographic characteristics may impact epigenetic factors which further contribute to this risk of gestational diabetes. The PRS generated through our study will be combined with an analysis of epigenetic factors to produce a new method for predicting risk of developing gestational diabetes during pregnancy.

DETAILED DESCRIPTION:
Gestational diabetes is a condition where high blood glucose levels occur during pregnancy and the mother was not diabetic before pregnancy. Between 6-9% of pregnancies are affected by this disorder. Gestational diabetes is usually diagnosed with a glucose challenge test where a blood glucose level of 190mg/dL or above would be indicative of gestational diabetes. This test usually occurs around 24-28 weeks into pregnancy. If a patient has other risk factors such as obesity or family history of diabetes, the assessment may be performed earlier.

Gestational diabetes increases risk of complications in both the mother and the baby. For the child, it may result in excessive weight at birth, a preterm birth, hypoglycemia, Type II diabetes later in life, and potential stillbirth. For the mother, it drastically increases the risk of high blood pressure, preeclampsia, and developing diabetes later in life. Gestational diabetes can also lead to further pregnancy related complications and increased risk of maternal morbidity and mortality events.

Very few genome-wide association studies have been carried out to correlate genetic variants to gestational diabetes, and have identified a small non-exhaustive number of genes linked to the condition. The list comprises genes encoding transcription factors such as TCF7L2 and genes required for glucose processing such as GCK and GCKR. Many of these genes are also associated with the risk of Type II diabetes. A large number of GWAS have identified genes tightly associated with Type II diabetes including CDKALI 1, FOXO1, GCKR and FTO, and the risk of gestational diabetes and type II is strongly correlated. These variants, along with demonstrated non-genetic risk factors such as obesity and high blood pressure, have demonstrated a clear ability to assess risk of different types of diabetes including gestational diabetes . However, there are currently no PRS for gestational diabetes available as a market product in any country. Additionally, the studies mentioned above do not wholly combine genome data with sociodemographic and lifestyle risks. Very few large scale GWAS studies have focused solely on female participants or pregnancy related complications. Further, existing literature and publications lack diversity among female participants and often focus on specific sub-populations. Prenome intends to conduct a large-scale GWAS in conjunction with the additional socioeconomic qualifications to generate a novel PRS to assess the risk of gestational diabetes with focus on inclusion of diverse populations in our samples. With these added quantifications of qualitative data, Prenome's PRS will be more representative of a patient's personal health and risk of developing gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females who are currently pregnant
* Adult females who have been pregnant within the last 12 months
* Adult female who is currently diagnosed with gestational diabetes
* Adult female who has been diagnosed with gestational diabetes within the last 12 months

Exclusion Criteria:

* Males
* Minors/ Children

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The population included in this study are pregnant or recently pregnant women, with a focus on women who are currently diagnosed or have previously been diagnosed with gestational diabetes. The population are being recruited from all adult age ranges, ethnicities, races and location across the united states.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Polygenic Risk Score Prediction for Gestational Diabetes | 1 year
  A predictive model of genetic risk of developing gestational diabetes based on comparing variants between control and diabetic groups.

SECONDARY OUTCOMES:
Impact of Social Determinants of Health on Risk | 1 year
  The impact of a social determinant from survey data on the generated genetic risk assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Levy, MD, Principal Investigator — Prenome
Locations (1):
- Illumina Accelerator, Foster City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Sign Up — https://www.prenome.com/clinical-study-oneinseven

DOCUMENTS (1):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT04789473/Prot_001.pdf